CLINICAL TRIAL: NCT01333683
Title: Tinnitus and Arterial Hypertension.is There Any Relationship?
Brief Title: Tinnitus and Arterial Hypertension
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Faculdade de Medicina de Valenca (Other)
Collaborators: Federal University of São Paulo (Other)
Responsible Party: Principal Investigator, Ricardo Rodrigues Figueiredo, M.D, MSc, Faculdade de Medicina de Valenca
Other Study IDs: HAS
Record Dates: First submitted 2011-04-07; First posted 2011-04-12 (Estimated); Last update posted 2015-03-06 (Estimated); Status verified 2015-03

CONDITIONS: Tinnitus; Hearing Loss; Arterial Hypertension
Keywords: tinnitus; hearing loss; arterial hypertension; ototoxicity
MeSH Terms: conditions — Tinnitus; Hearing Loss; Hypertension; Ototoxicity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Control: Normal subjects
- AH: Arterial hypertension patients

SUMMARY:
Many authors link tinnitus to arterial hypertension. The aim of this study is to establish a possible relationship between them, analyze the severity of tinnitus related to arterial hypertension and analyze a possible influence of ototoxic drugs used to treat arterial hypertension

DETAILED DESCRIPTION:
Arterial hypertension has been cited as a possible tinnitus etiology. Vascular abnormalities associated with it may account for cochlear and central nervous system. However, a relationship between tinnitus and arterial hypertension has never been established. The aim of this study is to analyze this relationship, comparing groups with and without arterial hypertension and the incidence of tinnitus amongst them. Inclusion and exclusion criteria try to isolate arterial hypertension as the main etiological factor, as much as possible. Presbycusis, noise exposure, metabolical diseases and genetic factors will be ruled out. A comparison will be performed inside the arterial hypertension group between subgroups that use or not ototoxic medications, such as furosemide and beta-blockers

ELIGIBILITY:
Inclusion Criteria:

* age between 40 and 50
* arterial hypertension for group 1
* at least 5 years standing arterial hypertension

Exclusion Criteria:

* chronic noise exposure
* metabolic diseases
* family antecedents of hearing loss (except for presbycusis)
* pregnant women
* use of ototoxic drugs (except for anti-hypertensives)

Ages: 40 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Patients agedd between 40 and 50
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2011-04; Primary Completion 2015-04 (Estimated); Study Completion 2015-10 (Estimated)

PRIMARY OUTCOMES:
Incidence of tinnitus - have tinnitus x don't have tinnitus | Up to 6 months
  The purpose of this study is to compare tinnitus incidence between patients with and without arterial hypertension.

SECONDARY OUTCOMES:
Severity of tinnitus - Tinnitus Handicap Inventory | Up to 6 months
  Severity of tinnitus measured by Tinnitus Handicap Inventory, to evaluate differences between patients with and without arterial hypertension

CONTACTS AND LOCATIONS:
Overall Officials: Ricardo R Figueiredo, MD,MSc, Principal Investigator — Otosul, Valença Medical School
Locations (1):
- Faculdade de Medicina de Valença, Valença, Rio de Janeiro, Brazil